CLINICAL TRIAL: NCT03382483
Title: A Prospective, Patient-centric, Observational, Consecutive Enrollment, Non-interventional Study of Patients At Risk for Fracture Non-union Treated With EXOGEN Compared to a National Healthcare Claims Database Control
Brief Title: Observational, Non-interventional Use of LIPUS to Mitigate Fracture Non-union in Patients at Risk
Acronym: BONES
Status: Completed | Type: Observational
Sponsor: Bioventus LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 16EXO401; 17EXO402 (Other: Bioventus); 17EXO403 (Other: Bioventus)
Record Dates: First submitted 2017-12-19; First posted 2017-12-26 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Mitigation of Fracture Non-union in Patients at Risk

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- EXOGEN Treated: Patients prescribed EXOGEN and treatment initiated
  Interventions: Device: Low intensity pulsed ultrasound
- Non-EXOGEN Treated: Patients in insurance claims database who have not been treated with a bone growth stimulator; derived via propensity score subclassification

INTERVENTIONS:
Device: Low intensity pulsed ultrasound — bone growth stimulator
  Other Names: EXOGEN
  Groups: EXOGEN Treated

SUMMARY:
This study is one of three separate studies of the Bioventus Observational Non-interventional EXOGEN Studies (BONES) program. Eligibility for each study is determined by fractured bone.

DETAILED DESCRIPTION:
The prospective arm of this non-interventional, observational study is designed to collect real world evidence from patients at risk of a fracture non-union across the US receiving EXOGEN treatment. Patients will be followed for 9 months post fracture. As a non-interventional study, the treating clinician will continue to provide routine care without research intervention or dictation by a protocol. A medically staffed Direct-to-Patient Contact Center will serve as a central investigational site with scheduled and structured direct-to-patient contacts via phone/email/text/web based surveys to obtain informed consent and collect data directly from the patient. For all prospective patients, primary effectiveness data will be obtained directly from the medical records of the treating physician.

The comparator arm of this study will be a retrospective cohort of patients within a national health insurance claims database. An extract of this database will be taken and eligible controls derived via propensity score analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Must be willing to provide voluntary informed consent
2. Male or female age 21-80 on fracture date
3. Must be willing to sign for release of medical insurance claim billing records from the treating clinician, pertaining to the fracture and fracture treatment
4. Fluency in English and/or Spanish
5. Prescriptive initiation of therapy with the EXOGEN Ultrasound Bone Healing System (Model number 71034400) for a specified fracture
6. Bone specific fracture

Exclusion Criteria:

1. Patient report of treatment with an electrical bone growth stimulation device (e.g., pulsed electromagnetic field (PEMF) or capacitive coupling (CC) based devices) for bone fracture in 9-months pre-index period up to baseline phone contact
2. Pregnant on fracture index date
3. Evidence that prescription for EXOGEN has been written to treat a fracture non-union or mal-union (i.e, ICD-10-CM code with seventh character modifier of K, P or S).
4. Evidence that prescription for EXOGEN has been written to treat a pathologic fracture (ICD-10-CM code M80. or M84.) or neuropathic bone (ICD-10-CM code M14.6)
5. Patient with a concurrent fracture of the other bones of interest
6. Patients who are or anticipate living or receiving fracture treatment outside of the US during the post-index fracture period
7. Patient report of history of primary or metastatic bone cancer
8. Patient report of bone infection or osteomyelitis of index fracture at baseline contact
9. Patient report of prior bone specific fracture in 9-months pre-index period
10. Patient prescribed EXOGEN as part of a Worker Compensation claim

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Prospective EXOGEN Treated Patients: Adult patients (21-80 years old) in the United States (US) at risk for the development of fracture non-union who have been prescribed EXOGEN as adjunctive treatment for a specific bone fracture.
  Retrospective Non-EXOGEN Treated Claims Data Cohort: Adult patients (21-80 years old) in the US at risk for development of fracture non-union who are covered under commercial insurance within the MarketScan database for 18 contiguous months.
Sampling Method: Probability Sample
Enrollment: 12387 (Actual)
Dates: Start 2017-10-16 (Actual); Primary Completion 2020-05-26 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Adjunctive treatment with low intensity pulsed ultrasound therapy mitigates the risk of fracture non-union in patients at risk | 9 month
  To compare incidence of fracture non-union in patients utilizing the EXOGEN device with patients receiving standard of care alone

CONTACTS AND LOCATIONS:
Overall Officials: Robert Zura, MD, Principal Investigator — LSU Head of Orthopedics; Christina Mack, PhD, MPH, Principal Investigator — IQUVIA
Locations (1):
- CliniCallRN, Jericho, New York, United States